CLINICAL TRIAL: NCT03031119
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess Safety, Tolerability, And Pharmacokinetics Of Multiple Oral Doses Of Pf-06835919 In Healthy Adult Subjects (Part A); And An Open-label Study To Assess Multiple Oral Doses Of Pf-06835919 On Atorvastatin Pharmacokinetics (Part B)
Brief Title: Multiple Ascending Dose and DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C1061002; 2016-004649-10 (EudraCT Number)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers
Keywords: nonalcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — PF-06835919; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Tablets administered once or twice daily, with food, in Part A for 14 days.
  Interventions: Drug: Placebo
- PF-06835919 (Experimental): Tablets administered once or twice daily, with food, in Part A for 14 days. Tablets administered once or twice daily, for 4 days at a low dose and for 4 days at a higher dose, with food and atorvastatin in Part B.
  Interventions: Drug: PF-06835919; Drug: atorvastatin
- atorvastatin (Experimental): In Part B, tablets administered once or twice daily, with food, with and without a low dose of PF-06835919 for 4 days and a higher dose of PF-06835919 for 4 days.
  Interventions: Drug: PF-06835919; Drug: atorvastatin

INTERVENTIONS:
Drug: Placebo — Tablets administered once or twice daily, with food, in Part A.
  Arms: Placebo
Drug: PF-06835919 — Tablets administered once or twice daily, with food, in Part A. Tablets administered once or twice daily, with food and atorvastatin in Part B.
  Arms: PF-06835919; atorvastatin
Drug: atorvastatin — In Part B, tablets administered once or twice daily, with food, with and without PF-06835919.
  Arms: PF-06835919; atorvastatin

SUMMARY:
Part A will investigate the safety, tolerability, PK and PD of PF-06835919 administered for 14 days in a multiple ascending dose design. Part B will assess the effect of PF-06835919 co-administration at low and high doses on the PK of atorvastatin in a single cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and females (nonchildbearing potential)
* 18 to 55 years old
* Body Mass Index 17.5 to 30.5

Exclusion Criteria:

* Known hereditary fructose intolerance or fructose malabsorption disorder (Part A)
* Statin intolerance (Part B)
* Unable to consume high fructose syrup-containing beverage with each meal while in the unit (Part A)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Screening to Day 24
  Part A
Number of Participants With Clinical Laboratory Abnormalities | Day -2 to Day 24
  Part A
Change from baseline in vital signs | Day -1 to Day 24
  Part A
Change from baseline in 12-lead electrocardiogram | Day -1 to Day 24
  Part A
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) on Day -1 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) on Day 3 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) on Day 7 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) on Day -1 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) on Day 3 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) on Day 7 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 3 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 7 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Maximum Observed Plasma Concentration (Cmax) on Day -1 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Maximum Observed Plasma Concentration (Cmax) on Day 3 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Maximum Observed Plasma Concentration (Cmax) on Day 7 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Plasma Decay Half-Life (t1/2) on Day -1 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Plasma Decay Half-Life (t1/2) on Day 3 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B
Plasma Decay Half-Life (t1/2) on Day 7 of atorvastatin and 2 active metabolites | 0,0.5,1,1.5,2,3,4,6,9,12,24,36 and 48 hours post-atorvastatin dose
  Part B

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) on Day 1 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Maximum Observed Plasma Concentration (Cmax) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Maximum Observed Plasma Concentration (Cmax) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48, and 72 hours post-dose
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) on Day 1 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Apparent Oral Clearance (CL/F) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Apparent Oral Clearance (CL/F) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Minimum Observed Plasma Trough Concentration (Cmin) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Minimum Observed Plasma Trough Concentration (Cmin) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Accumulation Ratio (Rac) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Accumulation Ratio (Rac) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Accumulation Ratio for Maximum Observed Plasma Concentration (Rac,Cmax) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose
Accumulation Ratio for Maximum Observed Plasma Concentration (Rac,Cmax) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Plasma Decay Half-Life (t1/2) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Apparent Volume of Distribution (Vz/F) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Cumulative Amount of Drug Recovered Unchanged in Urine (Ae) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Percent Cumulative Amount of Drug Recovered Unchanged in Urine (Ae%) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Renal Clearance (CLr) on Day 14 Part A | 0,0.5,1,2,4,5,6,8,12,14,16,24,36,48 and 72 hours post-dose
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Screening to Day 18
  Part B
Number of Participants With Clinical Laboratory Abnormalities | Day -2 to Day 18
  Part B
Change from Baseline in Vital Signs | Day -2 to Day 18
  Part B
Change from baseline in 12-lead electrocardiogram | Day -2 to Day 18
  Part B
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) on Day 7 Part A | 0,0.5,1,2,4,5,6,8 and 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1061002&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Multiple+Oral+Doses+Of+Pf-06835919+In+Healthy+Adult+Subjects+%28part+A%29%3B+And+An+Open-label+Study+To+Assess+Multiple+Oral+Doses+Of+Pf-06835919+On+Atorvastatin+Pharmacokinetics+%28part+B%29